CLINICAL TRIAL: NCT05430451
Title: Building Capacity and Promoting Smoking Cessation in the Community Via "Quit to Win" Contest 2022: Simple Physical Exercise With Instant Messaging Support for Smoking Cessation
Brief Title: Simple Physical Exercise With Instant Messaging Support for Smoking Via "Quit to Win" Contest 2022 (QTW2022)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Hong Kong Council on Smoking and Health (Other)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: QTW2022
Record Dates: First submitted 2022-06-16; First posted 2022-06-24 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Smoking Cessation
Keywords: Smoking cessation; Physical exercise; Instant messaging support; mHealth
MeSH Terms: conditions — Smoking Cessation; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief cessation advice (AWARD) + simple physical exercise with Instant Messaging (IM) support (Experimental): The integrated intervention of brief cessation advice (AWARD), and simple physical exercise practices with Instant Messaging (IM) support for craving management
  Interventions: Behavioral: AWARD advice; Behavioral: Referral card; Behavioral: Self-help smoking cessation booklet; Behavioral: Simple physical exercise training; Behavioral: Simple physical exercises with instant messaging support
- Brief cessation advice (AWARD) (Active Comparator): Brief cessation advice (AWARD)
  Interventions: Behavioral: AWARD advice; Behavioral: Referral card; Behavioral: Self-help smoking cessation booklet; Behavioral: SMS

INTERVENTIONS:
Behavioral: AWARD advice — Ask about smoking history, Warn about the high risk of smoking, Advise to quit as soon as possible, Refer to the smoking cessation services, and Do it again (if the smokers refused to set quit date).
Behavioral: Referral card — The content consists of brief information and highlights of existing smoking cessation services, contact methods, motivation information, and strong supporting messages or slogans.
Behavioral: Self-help smoking cessation booklet — The contents include information about the benefits of quitting, smoking and diseases, methods to quit, how to handle withdrawal symptoms, declaration of quitting, etc.
Behavioral: Simple physical exercise training — The simple exercises consist of a) Zero-time exercises (ZTEx), b) handgrip exercises, and c) resistance exercises. Participants will receive handgrips and elastic bands, and trained smoking cessation ambassadors will demonstrate and encourage the use of handgrip and elastic bands onsite with an instruction leaflet.
  Arms: Brief cessation advice (AWARD) + simple physical exercise with Instant Messaging (IM) support
Behavioral: Simple physical exercises with instant messaging support — During the 3-month instant messaging support, smoking cessation counselors will deliver regular messages to encourage the practices of simple physical exercise, provide strategies for managing craving and withdrawal symptoms, and provide information on smoking-related knowledge and available smoking cessation services. Our trained smoking cessation counselors will also provide real-time support upon participants' inquiries.
  Arms: Brief cessation advice (AWARD) + simple physical exercise with Instant Messaging (IM) support
Behavioral: SMS — SMS on follow-up survey reminders
  Arms: Brief cessation advice (AWARD)

SUMMARY:
This project aims to test the effectiveness of an integrated intervention of brief cessation advice (AWARD) and simple physical exercise with Instant Messaging (IM) support compared with control participants among current smokers who joined the contest.

DETAILED DESCRIPTION:
Although smoking prevalence is decreasing in Hong Kong, it accounts for over 7,000 deaths per year and a large amount of medical cost, long-term care, and productivity loss of US$ 688 million (0.6% Hong Kong GDP). Quitting is difficult because nicotine is highly addictive. Long-term habitual tobacco smoking could foster a series of physical and psychological dependence on nicotine, and thus induce cravings and nicotine withdrawal symptoms when remaining abstinent.

In addition to pharmacotherapy and behavioral counseling, exercise has shown promising effects on reducing craving, cigarette consumption, withdrawal symptoms, and increasing intention and attempt to quit. Randomized trials on smoking cessation have shown that vigorous or moderate exercise (including aerobics, brisk walking, and weightlifting) increases tobacco abstinence. However, these exercise-based smoking cessation trials were small-scaled with sample sizes ranging from 20 to 543, and mainly targeted the smokers who were motivated to quit (active treatment seekers). Most (15/20) of the vigorous or moderate exercises adopted in the smoking cessation trials required the participants to attend multiple exercise sessions (at least weekly for 5 months) under supervision or self-monitoring using equipment (e.g., pedometers) with a low proportion (<50%) of the participants achieved targeted level of attendance and exercise. The effects were short-term (end of treatment) and long-term (6 months or above) effects were uncertain, and cannot be generated in smokers who had low motivation to quit.

Mobile health (mHealth) is now a part of the World Health Organization's (WHO) strategies on combating smoking (http://www.who.int/tobacco/mhealth/en/) and has been used in many countries given its low cost and popular use. Instant messaging (IM) applications (apps) (e.g., WhatsApp, WeChat) are compatible with smartphones and allow sending interactive messages such as text, photos, video, animation, and files. The widespread availability of IM apps allows healthcare professionals to deliver health information and behavioral interventions through messaging. The QTW Contest 2017 using chat-based psychosocial support through IM apps effectively increased short-term (end of treatment, 3 months) and long-term (6 months since intervention initiation) smoking abstinence.

The chat-based IM support has the potential to support the use of other treatment components. The investigators aimed to test (1) the effectiveness of an integrated intervention of brief cessation advice (AWARD), simple physical exercise with Instant Messaging (IM) support compared with control participants among current smokers; (2) to explore participants' experience and perceptions towards the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents aged 18 or above
* Smoke at least 1 tobacco stick (includes HTP) per day or use e-cigarette daily in the preceding 3-month
* Able to communicate in Chinese (including reading Chinese in IM)
* Saliva cotinine 30 ng/ml or above
* Intent to quit / reduce smoking
* Able to use the instant messaging tool (e.g., WhatsApp, WeChat) for communication.

Exclusion Criteria:

* Smokers who have communication barriers (either physically or cognitively)
* Smokers who are currently participating in other SC programmes or services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1031 (Actual)
Dates: Start 2022-06-18 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Biochemically validated abstinence | 3-month follow-up
  Defined as exhaled CO level <4ppm and saliva cotinine level ≤30 ng/ml
Biochemically validated abstinence | 6-month follow-up
  Defined as exhaled CO level <4ppm and saliva cotinine level ≤30 ng/ml

SECONDARY OUTCOMES:
Physical exercise level | 3-month follow-up
  Measured by international physical activity questionnaire - short form (IPAQ-SF). The scale assesses the types and intensity of physical activity and sitting time that people do as part of their daily lives (during the last 7 days) are considered to estimate total physical activity in metabolic equivalent of task (MET)-min/week and time spent sitting.
Physical exercise level | 6-month follow-up
  Measured by international physical activity questionnaire - short form(IPAQ-SF). The scale assesses the types and intensity of physical activity and sitting time that people do as part of their daily lives (during the last 7 days) are considered to estimate total physical activity in metabolic equivalent of task (MET)-min/week and time spent sitting.
Smoking quit rate change from baseline at 3-month follow-up | 3-month follow-up
  Self-reported 7-day point prevalence (pp) quit rate at 3-month between the two groups
Smoking quit rate change from baseline at 6-month follow-up | 6-month follow-up
  Self-reported 7-day point prevalence (pp) quit rate at 6-month between the two groups
Smoking reduction rate change from baseline at 3-month follow-up | 3-month follow-up
  Rate of smoking reduction by at least half of baseline amount in the two groups
Smoking reduction rate change from baseline at 6-month follow-up | 6-month follow-up
  Rate of smoking reduction by at least half of baseline amount in the two groups
Intervention compliance at the end of treatment at 3 months follow-up | 3-month follow-up
  Rate of self-reported practice and frequency of simple physical exercise, IM engagement (replied for at least 2 messages confirmed by the conversation log)

CONTACTS AND LOCATIONS:
Overall Officials: Man Ping Wang, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Hong Kong Council on Smoking and Health (COSH), Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhao SZ, Li MY, Li YJ, Luk TT, Cheung DYT, Lai AYK, Tong HSC, Lai VWY, Lam TH, Wang MP. Mobile instant messaging supported brief physical exercise intervention for smoking cessation: a community-based, cluster randomised controlled trial. Thorax. 2026 Jan 23:thorax-2025-224130. doi: 10.1136/thorax-2025-224130. Online ahead of print. PMID 41513451